CLINICAL TRIAL: NCT03138512
Title: A Phase 3 Randomized, Double-Blind Study of Nivolumab Monotherapy or Nivolumab Combined With Ipilimumab vs Placebo in Participants With Localized Renal Cell Carcinoma Who Underwent Radical or Partial Nephrectomy and Who Are at High Risk of Relapse
Brief Title: A Study Comparing Nivolumab, Nivolumab in Combination With Ipilimumab and Placebo in Participants With Localized Kidney Cancer Who Underwent Surgery to Remove Part of a Kidney
Acronym: CheckMate 914
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA209-914; 2016-004502-34 (EudraCT Number)
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: localized; resected; adjuvant; Renal Cell Carcinoma; Kidney Cancer; Nephrectomy; Clear cell; High Risk of Relapse/Recurrence
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Recurrence | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A, Arm A: nivolumab + ipilimumab (Experimental)
  Interventions: Biological: nivolumab; Biological: ipilimumab
- Part A, Arm B: nivolumab placebo + ipilimumab placebo (Placebo Comparator)
  Interventions: Drug: nivolumab placebo; Drug: ipilimumab placebo
- Part B, Arm A: nivolumab + ipilimumab (Experimental)
  Interventions: Biological: nivolumab; Biological: ipilimumab
- Part B, Arm B: nivolumab placebo + ipilimumab placebo (Placebo Comparator)
  Interventions: Drug: nivolumab placebo; Drug: ipilimumab placebo
- Part B, Arm C: nivolumab + ipilimumab placebo (Experimental)
  Interventions: Biological: nivolumab; Drug: ipilimumab placebo

INTERVENTIONS:
Biological: nivolumab — Specified dose on specified days
  Other Names: Opdivo
  Arms: Part A, Arm A: nivolumab + ipilimumab; Part B, Arm A: nivolumab + ipilimumab; Part B, Arm C: nivolumab + ipilimumab placebo
Biological: ipilimumab — Specified dose on specified days
  Other Names: Yervoy
  Arms: Part A, Arm A: nivolumab + ipilimumab; Part B, Arm A: nivolumab + ipilimumab
Drug: nivolumab placebo — Specified dose on specified days
  Arms: Part A, Arm B: nivolumab placebo + ipilimumab placebo; Part B, Arm B: nivolumab placebo + ipilimumab placebo
Drug: ipilimumab placebo — Specified dose on specified days
  Arms: Part A, Arm B: nivolumab placebo + ipilimumab placebo; Part B, Arm B: nivolumab placebo + ipilimumab placebo; Part B, Arm C: nivolumab + ipilimumab placebo

SUMMARY:
The purpose of this study is to determine whether nivolmab alone or the combination of nivolumab and ipilimumab versus placebo, is safe and effective for delaying or preventing recurrence of cancer in participants who have experienced partial or entire removal of a kidney.

DETAILED DESCRIPTION:
The study has two primary endpoints. The first primary completion date is anticipated to be reached July 2022 (DFS in Part A). The second primary completion date is anticipated to be reached July 2024 (DFS in Part B).

ELIGIBILITY:
Inclusion Criteria:

* Kidney tumor has been completely resected with negative surgical margins obtained. The randomization must occur greater than 4 weeks and less than (or equal to) 12 weeks from the date of nephrectomy
* Pathologic tumor, node, and metastasis (TNM) staging meeting one of the following: pT2a, G3 or G4, N0 M0; pT2b, G any, N0 M0; pT3, (a, b, c), G any, N0 M0; pT4, G any, N0 M0; pT any, G any, N1 M0
* Post-nephrectomy tumor shows renal cell cancer (RCC) with a predominantly clear cell histology, including participants with sarcomatoid features
* Participants must have no clinical or radiological evidence of macroscopic residual disease or distant metastases after nephrectomy
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1
* Women must agree to follow methods of contraception, if applicable

Exclusion Criteria:

* Participants with an active known or suspected autoimmune disease
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Any severe or serious, acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation
* History of allergy or hypersensitivity to study drug components
* Participants with a condition requiring systemic treatment with corticosteroids
* Participants who have received a live/attenuated vaccine within 30 days of first treatment

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1641 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (200):
- United States (21):
  - Local Institution - 0019, Birmingham, Alabama
  - Local Institution - 0056, Springdale, Arkansas
  - Local Institution - 0186, Los Angeles, California
  - Local Institution - 0180, Los Angeles, California
  - Local Institution - 0002, San Francisco, California
  - Local Institution - 0185, Aurora, Colorado
  - Local Institution - 0016, Athens, Georgia
  - Local Institution - 0005, Chicago, Illinois
  - Local Institution, Chicago, Illinois
  - Local Institution - 0006, St Louis, Missouri
  - Local Institution - 0012, Howell Township, New Jersey
  - Local Institution - 0007, Buffalo, New York
  - Local Institution - 0181, New York, New York
  - Local Institution - 0001, New York, New York
  - Local Institution - 0008, Columbus, Ohio
  - Local Institution - 0009, Portland, Oregon
  - Local Institution - 0010, Allentown, Pennsylvania
  - Local Institution - 0014, Greenville, South Carolina
  - Local Institution - 0013, Chattanooga, Tennessee
  - Local Institution - 0183, Nashville, Tennessee
  - Local Institution - 0057, Fairfax, Virginia
- Argentina (13):
  - Local Institution - 0178, Capital Federal, Buenos Aires
  - Local Institution - 0126, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 0203, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0095, Mar del Plata, Buenos Aires
  - Local Institution - 0208, Mar del Plata, Buenos Aires
  - Local Institution - 0173, Río Cuarto, Córdoba Province
  - Local Institution - 0232, Bariloche, Río Negro Province
  - Local Institution - 0179, Buenos Aires
  - Local Institution - 0099, CABA
  - Local Institution - 0096, Córdoba
  - Local Institution - 0098, Córdoba
  - Local Institution - 0164, San Juan
  - Local Institution - 0097, San Miguel de Tucumán
- Australia (10):
  - Local Institution - 0215, Macquarie Park, New South Wales
  - Local Institution - 0032, Northmead, New South Wales
  - Local Institution - 0036, Randwick, New South Wales
  - Local Institution - 0035, St Leonards, New South Wales
  - Local Institution - 0113, South Brisbane, Queensland
  - Local Institution - 0213, Southport, Queensland
  - Local Institution - 0034, Elizabeth Vale, South Australia
  - Local Institution - 0033, Clayton, Victoria
  - Local Institution - 0214, Heidelberg, Victoria
  - Local Institution - 0031, Murdoch, Western Australia
- Austria (2):
  - Local Institution - 0068, Linz
  - Local Institution - 0084, Vienna
- Belgium (4):
  - Local Institution - 0058, Ghent, Oost-Vlaanderen
  - Local Institution - 0064, Anderlecht
  - Local Institution - 0060, Hasselt
  - Local Institution - 0059, Liège
- Brazil (8):
  - Local Institution - 0047, Brasília, Federal District
  - Local Institution - 0045, Belo Horizonte, Minas Gerais
  - Local Institution - 0046, Ijuí, Rio Grande do Sul
  - Local Institution - 0048, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0043, Barretos, São Paulo
  - Local Institution - 0044, São Paulo, São Paulo
  - Local Institution - 0160, Rio de Janeiro
  - Local Institution - 0050, São Paulo
- Canada (6):
  - Local Institution - 0041, Vancouver, British Columbia
  - Local Institution - 0086, Saint John, New Brunswick
  - Local Institution - 0087, Oshawa, Ontario
  - Local Institution - 0112, Toronto, Ontario
  - Local Institution - 0042, Montreal, Quebec
  - Local Institution - 0040, Rimouski, Quebec
- Chile (5):
  - Local Institution - 0223, La Serena, Coquimbo Region
  - Local Institution - 0222, Viña del Mar, Región de Valparaíso
  - Local Institution - 0246, Santiago, Santiago Metropolitan
  - Local Institution, Santiago, Santiago Metropolitan
  - Local Institution - 0221, Santiago, Santiago Metropolitan
- China (24):
  - Local Institution - 0147, Beijing, Beijing Municipality
  - Local Institution - 0153, Beijing, Beijing Municipality
  - Local Institution - 0159, Beijing, Beijing Municipality
  - Local Institution - 0132, Fuzhou, Fujian
  - Local Institution - 0141, Guangzhou, Guangdong
  - Local Institution - 0194, Wuhan, Hebei
  - Local Institution - 0133, Wuhan, Hubei
  - Local Institution - 0138, Nanjing, Jiangsu
  - Local Institution - 0140, Nanchang, Jiangxi
  - Local Institution - 0145, Changchun, Jilin
  - Local Institution - 0144, Xi'an, Shan3xi
  - Local Institution - 0146, Yantai, Shandong
  - Local Institution - 0137, Shanghai, Shanghai Municipality
  - Local Institution - 0166, Shanghai, Shanghai Municipality
  - Local Institution - 0152, Shanghai, Shanghai Municipality
  - Local Institution - 0148, Shanghai, Shanghai Municipality
  - Local Institution - 0142, Chengdu, Sichuan
  - Local Institution - 0143, Chengdu, Sichuan
  - Local Institution - 0175, Tianjin, Tianjin Municipality
  - Local Institution - 0157, Hangzhou, Zhejiang
  - Local Institution - 0131, Hangzhou, Zhejiang
  - Local Institution - 0134, Guangzhou
  - Local Institution - 0139, Nanjing
  - Local Institution - 0176, Shanghai
- Colombia (5):
  - Local Institution - 0227, Medellín, Antioquia
  - Local Institution - 0228, Valledupar, Cesar Department
  - Local Institution - 0229, Bogotá
  - Local Institution - 0230, Floridablanca
  - Local Institution - 0226, Pereira
- Czechia (2):
  - Local Institution - 0094, Hradec Králové
  - Local Institution - 0025, Olomouc
- France (12):
  - Local Institution - 0083, Besançon
  - Local Institution - 0080, Bordeaux
  - Local Institution - 0082, La Roche-sur-Yon
  - Local Institution - 0116, Lyon
  - Local Institution - 0079, Marseille
  - Local Institution - 0198, Paris
  - Local Institution - 0081, Rennes
  - Local Institution - 0077, Strasbourg
  - Local Institution - 0115, Toulouse
  - Local Institution - 0150, Tours
  - Local Institution - 0078, Vandœuvre-lès-Nancy
  - Local Institution - 0076, Villejuif
- Germany (11):
  - Local Institution - 0217, Tübingen, Baden-Wurttemberg
  - Local Institution - 0053, Aachen
  - Local Institution - 0103, Essen
  - Local Institution - 0052, Hamburg
  - Local Institution - 0231, Hanover
  - Local Institution - 0061, Hanover
  - Local Institution - 0062, Jena
  - Local Institution - 0102, Munich
  - Local Institution - 0054, Nuremberg
  - Local Institution - 0055, Rostock
  - Local Institution - 0101, Würzburg
- Italy (6):
  - Local Institution - 0105, Arezzo
  - Local Institution - 0172, Cremona
  - Local Institution - 0106, Napoli
  - Local Institution - 0107, Parma
  - Local Institution - 0109, Roma
  - Local Institution - 0108, Verona
- Japan (24):
  - Local Institution - 0129, Toyoake Shi, Aichi-ken
  - Local Institution - 0193, Hirosaki-shi, Aomori
  - Local Institution - 0158, Chiba, Chiba
  - Local Institution - 0121, Fukuoka, Fukuoka
  - Local Institution - 0156, Sapporo, Hokkaido
  - Local Institution - 0167, Kobe, Hyōgo
  - Local Institution - 0191, Tsukuba, Ibaraki
  - Local Institution - 0168, Shiwa-gun, Iwate
  - Local Institution - 0128, Yokohama, Kanagawa
  - Local Institution - 0216, Kumamoto, Kumamoto
  - Local Institution - 0130, Kamigyō-ku, Kyoto
  - Local Institution - 0123, Nagasaki, Nagasaki
  - Local Institution - 0120, Niigata, Niigata
  - Local Institution - 0125, Osakasayama-shi, Osaka
  - Local Institution - 0122, Suita-shi, Osaka
  - Local Institution - 0162, Tokushima, Tokushima
  - Local Institution - 0188, Adachi-ku, Tokyo
  - Local Institution - 0189, Bunkyo-ku, Tokyo
  - Local Institution - 0119, Bunkyo-ku, Tokyo
  - Local Institution - 0149, Shinjuku-ku, Tokyo
  - Local Institution - 0163, Ube-shi, Yamaguchi
  - Local Institution - 0165, Hiroshima
  - Local Institution - 0192, Wakayama
  - Local Institution - 0127, Yamagata
- Mexico (11):
  - Local Institution - 0197, Tuxtla Gutiérrez, Chiapas
  - Local Institution - 0195, Torreón, Coahuila
  - Local Institution - 0242, Tijuana, Estado de Baja California
  - Local Institution - 0110, Zapopan, Jalisco
  - Local Institution - 0151, Mexico City, Mexico City
  - Local Institution - 0111, Tlalpan, Mexico City
  - Local Institution - 0104, Mazatlán, Sinaloa
  - Local Institution - 0196, Mérida, Yucatán
  - Local Institution - 0089, Chihuahua City
  - Local Institution - 0088, Monterrey, NL
  - Local Institution - 0169, San Luis Potosí City
- Netherlands (3):
  - Local Institution - 0066, Amsterdam
  - Local Institution - 0067, Rotterdam
  - Local Institution - 0092, Zwolle
- Poland (2):
  - Local Institution - 0155, Bydgoszcz
  - Local Institution - 0038, Wroclaw
- Romania (5):
  - Local Institution - 0243, Bucharest
  - Local Institution - 0200, Cluj-Napoca
  - Local Institution - 0247, Cluj-Napoca
  - Local Institution - 0199, Craiova
  - Local Institution - 0202, Iași
- Russia (4):
  - Local Institution - 0065, Moscow
  - Local Institution - 0170, Novosibirsk
  - Local Institution - 0171, Saint Petersburg
  - Local Institution - 0021, Saint Petersburg
- Singapore (2):
  - Local Institution - 0018, Singapore, Central Singapore
  - Local Institution - 0017, Singapore
- Spain (9):
  - Local Institution - 0204, Barcelona
  - Local Institution - 0206, Barcelona
  - Local Institution - 0124, Cáceres
  - Local Institution - 0207, Córdoba
  - Local Institution - 0118, Lugo
  - Local Institution - 0114, Madrid
  - Local Institution - 0205, Madrid
  - Local Institution - 0117, Sabadell
  - Local Institution - 0161, Seville
- Switzerland (3):
  - Local Institution - 0218, Chur
  - Local Institution - 0219, Sankt Gallen
  - Local Institution - 0225, Zurich
- Turkey (Türkiye) (3):
  - Local Institution - 0209, Ankara
  - Local Institution - 0210, Istanbul
  - Local Institution, Istanbul
- United Kingdom (5):
  - Local Institution - 0075, Southampton, Hampshire
  - Local Institution - 0063, Manchester
  - Local Institution - 0071, Northwood
  - Local Institution - 0073, Preston
  - Local Institution - 0072, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Motzer RJ, Bex A, Russo P, Tomita Y, Cutuli HJ, Rojas C, Gross-Goupil M, Schinzari G, Melichar B, Barthelemy P, Ruiz Garcia A, Sosman J, Grimm MO, Goh JC, Suarez C, Kollmannsberger CK, Nair SG, Shuch BM, Huang J, Simsek B, Spiridigliozzi J, Lee CW, van Kooten Losio M, Grunwald V. Adjuvant Nivolumab for Localized Renal Cell Carcinoma at High Risk of Recurrence After Nephrectomy: Part B of the Randomized, Placebo-Controlled, Phase III CheckMate 914 Trial. J Clin Oncol. 2025 Jan 10;43(2):189-200. doi: 10.1200/JCO.24.00773. Epub 2024 Sep 20. PMID 39303200
- [Derived] Motzer RJ, Russo P, Grunwald V, Tomita Y, Zurawski B, Parikh O, Buti S, Barthelemy P, Goh JC, Ye D, Lingua A, Lattouf JB, Albiges L, George S, Shuch B, Sosman J, Staehler M, Vazquez Estevez S, Simsek B, Spiridigliozzi J, Chudnovsky A, Bex A. Adjuvant nivolumab plus ipilimumab versus placebo for localised renal cell carcinoma after nephrectomy (CheckMate 914): a double-blind, randomised, phase 3 trial. Lancet. 2023 Mar 11;401(10379):821-832. doi: 10.1016/S0140-6736(22)02574-0. Epub 2023 Feb 9. PMID 36774933
- [Derived] Marconi L, Sun M, Beisland C, Klatte T, Ljungberg B, Stewart GD, Dabestani S, Choueiri TK, Bex A. Prevalence, Disease-free, and Overall Survival of Contemporary Patients With Renal Cell Carcinoma Eligible for Adjuvant Checkpoint Inhibitor Trials. Clin Genitourin Cancer. 2021 Apr;19(2):e92-e99. doi: 10.1016/j.clgc.2020.12.005. Epub 2021 Jan 7. PMID 33526329
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A and B participants are separately randomized and treated.
Groups:
- Treatment Part A: Nivo + Ipi; Treatment Part B: Nivo + Ipi: Nivolumab 240 mg every 2 weeks and ipilimumab 1 mg/kg every 6 weeks (or every third nivolumab dose if dosing is delayed).
- Treatment Part A: Placebo; Treatment Part B: Placebo: Placebo infusions at the same frequency of nivolumab and ipilimumab infusions.
- Treatment Part B: Nivo: Nivolumab 240 mg every 2 weeks and ipilimumab Placebo every 6 weeks (or every third nivolumab dose if dosing is delayed).
Period: Randomization
Arm/Group | Treatment Part A: Nivo + Ipi | Treatment Part A: Placebo | Treatment Part B: Nivo + Ipi | Treatment Part B: Placebo | Treatment Part B: Nivo
Started | 405 | 411 | 206 | 208 | 411
Completed (Continuing to Treatment) | 404 | 407 | 204 | 207 | 408
Not Completed | 1 | 4 | 2 | 1 | 3
Not completed — Participants withdrew consent | 0 | 1 | 1 | 0 | 0
Not completed — Participant no longer meets study criteria | 0 | 3 | 1 | 1 | 3
Not completed — Other reasons | 1 | 0 | 0 | 0 | 0
Period: Treatment Part A
Arm/Group | Treatment Part A: Nivo + Ipi | Treatment Part A: Placebo | Treatment Part B: Nivo + Ipi | Treatment Part B: Placebo | Treatment Part B: Nivo
Started | 404 | 407 | 0 | 0 | 0
Completed | 229 | 360 | 0 | 0 | 0
Not Completed | 175 | 47 | 0 | 0 | 0
Not completed — Disease recurrence | 10 | 20 | 0 | 0 | 0
Not completed — Study Drug Toxicity | 132 | 5 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Adverse event unrelated to study drug | 9 | 4 | 0 | 0 | 0
Not completed — Participant request to discontinue treatment | 9 | 4 | 0 | 0 | 0
Not completed — Participant withdrew consent | 2 | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Poor/non-compliance | 1 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0
Not completed — Other reasons | 11 | 8 | 0 | 0 | 0
Period: Treatment Part B
Arm/Group | Treatment Part A: Nivo + Ipi | Treatment Part A: Placebo | Treatment Part B: Nivo + Ipi | Treatment Part B: Placebo | Treatment Part B: Nivo
Started | 0 | 0 | 204 | 207 | 408
Completed | 0 | 0 | 118 | 182 | 327
Not Completed | 0 | 0 | 86 | 25 | 81
Not completed — Disease recurrence | 0 | 0 | 6 | 12 | 10
Not completed — Study drug toxicity | 0 | 0 | 63 | 3 | 45
Not completed — Death | 0 | 0 | 1 | 0 | 0
Not completed — Adverse event unrelated to study drug | 0 | 0 | 5 | 2 | 12
Not completed — Participants request to discontinue study treatment | 0 | 0 | 6 | 4 | 6
Not completed — Participant withdrew consent | 0 | 0 | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Poor/non-compliance | 0 | 0 | 1 | 1 | 1
Not completed — Other reasons | 0 | 0 | 3 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Part A: Nivo + Ipi | Treatment Part A: Placebo | Treatment Part B: Nivo + Ipi | Treatment Part B: Placebo | Treatment Part B: Nivo | Total
Number analyzed (Participants) | 405 | 411 | 206 | 208 | 411 | 1641
Age, Customized [Count of Participants; unit: Participants] — Population: Part A and B are separately treated participants. The combined number of participants from Part A and B are equal to the total number randomized to this study.
  Participants
    < 65 | 293 | 301 | 132 | 137 | 279 | 1142
    >= 65 AND < 75 | 93 | 91 | 64 | 60 | 108 | 416
    >= 75 AND < 85 | 19 | 19 | 10 | 11 | 23 | 82
    >= 85 | 0 | 0 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Part A and B are separately treated participants. The combined number of participants from Part A and B are equal to the total number randomized to this study.
  Participants
    Female | 119 | 117 | 59 | 67 | 106 | 468
    Male | 286 | 294 | 147 | 141 | 305 | 1173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Part A and B are separately treated participants. The combined number of participants from Part A and B are equal to the total number randomized to this study.
  Participants
    Hispanic or Latino | 41 | 44 | 26 | 34 | 67 | 212
    Not Hispanic or Latino | 189 | 197 | 93 | 79 | 157 | 715
    Unknown or Not Reported | 175 | 170 | 87 | 95 | 187 | 714
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Part A and B are separately treated participants. The combined number of participants from Part A and B are equal to the total number randomized to this study.
  Participants
    American Indian or Alaska Native | 0 | 3 | 5 | 3 | 14 | 25
    Asian | 93 | 65 | 20 | 26 | 50 | 254
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 1
    Black or African American | 3 | 6 | 0 | 1 | 4 | 14
    White | 303 | 322 | 173 | 169 | 331 | 1298
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 6 | 14 | 8 | 9 | 12 | 49

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival (DFS) by BICR - Treatment Part A and B
Description: Disease-Free Survival (DFS) is defined as the time from randomization to development of local disease recurrence (ie, recurrence of primary tumor in situ or occurrence of a secondary renal cell carcinoma (RCC) primary cancer), distance metastasis, or death, whichever came first per Blinded Independent Central Review (BICR) based on Kaplan-Meier estimates.
Time Frame: From randomization to development of local disease recurrence, distance metastasis, or death, whichever came first (up to approximately 72 months)
Population: All randomized participants in Treatment Part A (Nivo + Ipi and Placebo Arms) and Treatment Part B (Placebo and Nivo Arms). The Nivo + Ipi Arm was prespecified to be excluded from the endpoint objective for Treatment Part B.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Part A: Nivo + Ipi | Treatment Part A: Placebo | Treatment Part B: Nivo + Ipi | Treatment Part B: Placebo | Treatment Part B: Nivo
Number analyzed (Participants) | 405 | 411 | 0 | 208 | 411
Months | NA [NA to NA] — Insufficient number of participants with events | NA [65.58 to NA] — Insufficient number of participants with events |  | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Treatment Part A: Nivo + Ipi vs Treatment Part A: Placebo; Test type: Superiority; p = 0.6676, Log Rank; Cox Proportional Hazard = 0.95, 95% CI [0.75 to 1.20]
Statistical Analysis 2: Comparison: Treatment Part A: Placebo vs Treatment Part B: Nivo; Test type: Superiority; p = 0.6556, Log Rank; Cox Proportional Hazard = 0.93, 95% CI [0.67 to 1.28]

2. Secondary Outcome: Overall Survival (OS) - Treatment Part A and B
Description: Overall Survival (OS) is defined as the time between the date of randomization and the date of death. For participants without documentation of death, OS will be censored on the last date the participants was known to be alive. Based on Kaplan-Meier estimates.
Time Frame: From randomization to the date of death (up to approximately 72 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Part A: Nivo + Ipi | Treatment Part A: Placebo | Treatment Part B: Nivo + Ipi | Treatment Part B: Placebo | Treatment Part B: Nivo
Number analyzed (Participants) | 405 | 411 | 0 | 208 | 411
Months | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events |  | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Treatment Part A: Nivo + Ipi vs Treatment Part A: Placebo; Treatment Part A; Test type: Superiority; p = 0.2436, Log Rank; Cox Proportional Hazard = 1.26, 95% CI [0.85 to 1.85]
Statistical Analysis 2: Comparison: Treatment Part A: Placebo vs Treatment Part B: Nivo; Treatment Part B; Test type: Superiority; p = 0.4500, Log Rank; Cox Proportional Hazard = 1.36, 95% CI [0.61 to 3.07]

3. Secondary Outcome: Overall Survival (OS) Rate (5 Years) - Treatment Part A and B
Description: Overall survival rate at 5 years is defined as the percentage of participants who are alive at 5 years.
Time Frame: At 5 years
Population: All randomized participants in Treatment Part A (Nivo + Ipi and Placebo Arms). Data was not collected for Treatment Part B.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Treatment Part A: Nivo + Ipi | Treatment Part A: Placebo | Treatment Part B: Nivo + Ipi | Treatment Part B: Placebo | Treatment Part B: Nivo
Number analyzed (Participants) | 405 | 411 | 0 | 0 | 0
Percent of participants | 85.0 [80.8 to 88.3] | 87.2 [82.8 to 90.5] |  |  |

4. Secondary Outcome: Disease-Free Survival (DFS) Per BICR in Contemporaneously Randomized Combination and Monotherapy Participants - Treatment Part B
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All randomized Nivo + Ipi and Nivo participants in Treatment Part B. Prespecified to be collected for Treatment Part B only. The Placebo Arm was prespecified to be excluded from the endpoint objective.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Part B: Nivo + Ipi | Treatment Part B: Nivo
Number analyzed (Participants) | 206 | 411
Months | NA [36.17 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Treatment Part B: Nivo + Ipi vs Treatment Part B: Nivo; Test type: Superiority; Cox Proportional Hazard = 1.22, 95% CI 2-sided [0.89 to 1.67]

5. Secondary Outcome: Overall Survival (OS) in the Contemporaneously Randomized Combination and Monotherapy Participants - Treatment Part B
Description: as for outcome 2
Time Frame: From randomization to the date of death (up to approximately 72 months)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Part B: Nivo + Ipi | Treatment Part B: Nivo
Number analyzed (Participants) | 206 | 411
Months | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Treatment Part B: Nivo + Ipi vs Treatment Part B: Nivo; Test type: Superiority; Cox Proportional Hazard = 0.75, 95% CI [0.33 to 1.68]

6. Secondary Outcome: The Number of Participants With Adverse Events up to 30 Days After Last Dose of Study Therapy - Treatment Part A
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Graded according to NCI CTCAE (Version 4) guidelines where grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life threatening, grade 5 = death.
Time Frame: From first dose to 30 days post last dose (up to approximately 40 weeks)
Population: All Treated Participants in Treatment Part A
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Part A: Nivo + Ipi | Treatment Part A: Placebo
Number analyzed (Participants) | 404 | 407
Participants
  Any Grade AE | 392 | 362
  Grade 3-4 AE | 154 | 44
  Grade 5 AE | 1 | 0
  Any Grade Drug-Related AE | 359 | 230
  Grade 3-4 Drug-Related AE | 114 | 8
  Grade 5 Drug-Related AE | 0 | 0

7. Secondary Outcome: The Number of Participants With Adverse Events up to 30 Days After Last Dose of Study Therapy - Treatment Part B
Description: as for outcome 6
Time Frame: From first dose to 30 days post last dose (up to approximately 40 weeks)
Population: All Treated Participants in Treatment Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Part B: Nivo + Ipi | Treatment Part B: Placebo | Treatment Part B: Nivo
Number analyzed (Participants) | 204 | 207 | 408
Participants
  Any Grade AE | 193 | 182 | 362
  Grade 3-4 AE | 59 | 31 | 70
  Grade 5 AE | 1 | 1 | 0
  Any Grade Drug-Related AE | 173 | 107 | 297
  Grade 3-4 Drug-Related AE | 41 | 4 | 36
  Grade 5 Drug-Related AE | 0 | 0 | 0

8. Secondary Outcome: The Number of Participants With Adverse Events up to 100 Days After Last Dose of Study Therapy - Treatment Part A
Description: as for outcome 6
Time Frame: From first dose to 100 days post last dose (up to approximately 50 weeks)
Population: All Treated Participants in Treatment Part A
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Part A: Nivo + Ipi | Treatment Part A: Placebo
Number analyzed (Participants) | 404 | 407
Participants
  Any Grade AE | 393 | 365
  Grade 3-4 AE | 167 | 52
  Grade 5 AE | 4 | 1
  Any Grade Drug-Related AE | 361 | 230
  Grade 3-4 Drug-Related AE | 128 | 9
  Grade 5 Drug-Related AE | 2 | 0

9. Secondary Outcome: The Number of Participants With Adverse Events up to 100 Days After Last Dose of Study Therapy - Treatment Part B
Description: as for outcome 6
Time Frame: From first dose to 100 days post last dose (up to approximately 50 weeks)
Population: All Treated Participants in Treatment Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Part B: Nivo + Ipi | Treatment Part B: Placebo | Treatment Part B: Nivo
Number analyzed (Participants) | 204 | 207 | 408
Participants
  Any Grade AE | 196 | 182 | 367
  Grade 3-4 AE | 68 | 32 | 85
  Grade 5 AE | 5 | 2 | 2
  Any Grade Drug-Related AE | 175 | 108 | 300
  Grade 3-4 Drug-Related AE | 46 | 5 | 46
  Grade 5 Drug-Related AE | 0 | 0 | 0

10. Secondary Outcome: The Number of Participants Experiencing Laboratory Parameters by Worst CTC (Grade 3-4) That Worsened Relative to Baseline up to 30 Days - Treatment Part A
Description: Graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE, Version 4.0] where grade 3 = severe, and grade 4 = life-threatening. Baseline evaluations are defined as evaluations or events that occur before the date and time of the first dose of study treatment.
Time Frame: From first dose to 30 days post last dose (up to approximately 40 weeks)
Population: All treated participants in Treatment Part A with a CTC graded laboratory result for the given parameter from both baseline and on-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Part A: Nivo + Ipi | Treatment Part A: Placebo
Number analyzed (Participants) | 398 | 404
Participants
  HEMOGLOBIN | 1 | 1
  PLATELET COUNT | 1 | 0
  LEUKOCYTES, LOCAL LAB | 0 | 0
  LYMPHOCYTES (ABSOLUTE), TOTAL | 6 | 3
  ABSOLUTE NEUTROPHIL COUNT | 2 | 0
  ALKALINE PHOSPHATASE, LOCAL LAB: number analyzed (Participants) | 397 | 404
  ALKALINE PHOSPHATASE, LOCAL LAB | 3 | 0
  ASPARTATE AMINOTRANSFERASE, LOCAL LAB | 14 | 3
  ALANINE AMINOTRANSFERASE, LOCAL LAB | 16 | 5
  BILIRUBIN, TOTAL, LOCAL LAB: number analyzed (Participants) | 395 | 404
  BILIRUBIN, TOTAL, LOCAL LAB | 1 | 0
  CREATININE, LOCAL LAB | 1 | 1
  HYPERNATREMIA | 0 | 0
  HYPONATREMIA | 28 | 7
  HYPERKALEMIA | 6 | 5
  HYPOKALEMIA | 3 | 1
  HYPERCALCEMIA: number analyzed (Participants) | 381 | 389
  HYPERCALCEMIA | 3 | 0
  HYPOCALCEMIA: number analyzed (Participants) | 381 | 389
  HYPOCALCEMIA | 1 | 0
  HYPERMAGNESEMIA: number analyzed (Participants) | 392 | 401
  HYPERMAGNESEMIA | 1 | 1
  HYPOMAGNESEMIA: number analyzed (Participants) | 392 | 401
  HYPOMAGNESEMIA | 1 | 0
  HYPERGLYCEMIA: number analyzed (Participants) | 180 | 179
  HYPERGLYCEMIA | 6 | 1
  HYPOGLYCEMIA: number analyzed (Participants) | 391 | 397
  HYPOGLYCEMIA | 1 | 0

11. Secondary Outcome: The Number of Participants Experiencing Laboratory Parameters by Worst CTC (Grade 3-4) That Worsened Relative to Baseline up to 30 Days - Treatment Part B
Description: as for outcome 10
Time Frame: From first dose to 30 days post last dose (up to approximately 40 weeks)
Population: All treated participants in Treatment Part B with a CTC graded laboratory result for the given parameter from both baseline and on-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Part B: Nivo + Ipi | Treatment Part B: Placebo | Treatment Part B: Nivo
Number analyzed (Participants) | 201 | 205 | 406
Participants
  HEMOGLOBIN | 0 | 3 | 0
  PLATELET COUNT: number analyzed (Participants) | 201 | 204 | 406
  PLATELET COUNT | 0 | 1 | 0
  LEUKOCYTES, LOCAL LAB | 0 | 0 | 1
  LYMPHOCYTES (ABSOLUTE), TOTAL | 3 | 1 | 4
  ABSOLUTE NEUTROPHIL COUNT | 0 | 0 | 1
  ALKALINE PHOSPHATASE, LOCAL LAB: number analyzed (Participants) | 201 | 205 | 404
  ALKALINE PHOSPHATASE, LOCAL LAB | 1 | 1 | 0
  ASPARTATE AMINOTRANSFERASE, LOCAL LAB: number analyzed (Participants) | 201 | 205 | 405
  ASPARTATE AMINOTRANSFERASE, LOCAL LAB | 4 | 4 | 5
  ALANINE AMINOTRANSFERASE, LOCAL LAB: number analyzed (Participants) | 201 | 205 | 405
  ALANINE AMINOTRANSFERASE, LOCAL LAB | 7 | 3 | 8
  BILIRUBIN, TOTAL, LOCAL LAB: number analyzed (Participants) | 200 | 205 | 405
  BILIRUBIN, TOTAL, LOCAL LAB | 0 | 1 | 0
  CREATININE, LOCAL LAB | 3 | 0 | 0
  HYPERNATREMIA: number analyzed (Participants) | 201 | 204 | 405
  HYPERNATREMIA | 0 | 0 | 0
  HYPONATREMIA: number analyzed (Participants) | 201 | 204 | 405
  HYPONATREMIA | 11 | 1 | 9
  HYPERKALEMIA | 1 | 2 | 2
  HYPOKALEMIA | 1 | 1 | 0
  HYPERCALCEMIA: number analyzed (Participants) | 197 | 199 | 396
  HYPERCALCEMIA | 1 | 0 | 1
  HYPOCALCEMIA: number analyzed (Participants) | 197 | 199 | 396
  HYPOCALCEMIA | 0 | 1 | 0
  HYPERMAGNESEMIA: number analyzed (Participants) | 196 | 203 | 404
  HYPERMAGNESEMIA | 2 | 2 | 3
  HYPOMAGNESEMIA: number analyzed (Participants) | 196 | 203 | 404
  HYPOMAGNESEMIA | 0 | 1 | 1
  HYPERGLYCEMIA: number analyzed (Participants) | 99 | 109 | 208
  HYPERGLYCEMIA | 3 | 1 | 3
  HYPOGLYCEMIA: number analyzed (Participants) | 196 | 195 | 401
  HYPOGLYCEMIA | 0 | 0 | 1

12. Secondary Outcome: The Number of Participants Experiencing Laboratory Parameters by Worst CTC (Grade 3-4) That Worsened Relative to Baseline up to 100 Days - Treatment Part A
Description: as for outcome 10
Time Frame: From first dose to 100 days post last dose (up to approximately 50 weeks)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Part A: Nivo + Ipi | Treatment Part A: Placebo
Number analyzed (Participants) | 401 | 406
Participants
  HEMOGLOBIN | 1 | 1
  PLATELET COUNT | 1 | 0
  LEUKOCYTES, LOCAL LAB | 0 | 0
  LYMPHOCYTES (ABSOLUTE), TOTAL | 11 | 3
  ABSOLUTE NEUTROPHIL COUNT | 2 | 0
  ALKALINE PHOSPHATASE, LOCAL LAB: number analyzed (Participants) | 400 | 406
  ALKALINE PHOSPHATASE, LOCAL LAB | 5 | 0
  ASPARTATE AMINOTRANSFERASE, LOCAL LAB | 17 | 3
  ALANINE AMINOTRANSFERASE, LOCAL LAB | 20 | 6
  BILIRUBIN, TOTAL, LOCAL LAB: number analyzed (Participants) | 399 | 406
  BILIRUBIN, TOTAL, LOCAL LAB | 3 | 0
  CREATININE, LOCAL LAB | 4 | 1
  HYPERNATREMIA | 0 | 0
  HYPONATREMIA | 30 | 7
  HYPERKALEMIA | 6 | 5
  HYPOKALEMIA | 5 | 1
  HYPERCALCEMIA: number analyzed (Participants) | 384 | 391
  HYPERCALCEMIA | 3 | 0
  HYPOCALCEMIA: number analyzed (Participants) | 384 | 391
  HYPOCALCEMIA | 1 | 0
  HYPERMAGNESEMIA: number analyzed (Participants) | 395 | 403
  HYPERMAGNESEMIA | 1 | 1
  HYPOMAGNESEMIA: number analyzed (Participants) | 395 | 403
  HYPOMAGNESEMIA | 1 | 0
  HYPERGLYCEMIA: number analyzed (Participants) | 183 | 179
  HYPERGLYCEMIA | 7 | 1
  HYPOGLYCEMIA: number analyzed (Participants) | 394 | 398
  HYPOGLYCEMIA | 1 | 0

13. Secondary Outcome: The Number of Participants Experiencing Laboratory Parameters by Worst CTC (Grade 3-4) That Worsened Relative to Baseline up to 100 Days - Treatment Part B
Description: as for outcome 10
Time Frame: From first dose to 100 days post last dose (up to approximately 50 weeks)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Part B: Nivo + Ipi | Treatment Part B: Placebo | Treatment Part B: Nivo
Number analyzed (Participants) | 203 | 205 | 407
Participants
  HEMOGLOBIN | 2 | 3 | 1
  PLATELET COUNT: number analyzed (Participants) | 203 | 204 | 407
  PLATELET COUNT | 0 | 1 | 0
  LEUKOCYTES, LOCAL LAB | 0 | 0 | 2
  LYMPHOCYTES (ABSOLUTE), TOTAL | 3 | 2 | 7
  ABSOLUTE NEUTROPHIL COUNT | 0 | 0 | 2
  ALKALINE PHOSPHATASE, LOCAL LAB: number analyzed (Participants) | 203 | 205 | 405
  ALKALINE PHOSPHATASE, LOCAL LAB | 2 | 1 | 0
  ASPARTATE AMINOTRANSFERASE, LOCAL LAB: number analyzed (Participants) | 203 | 205 | 406
  ASPARTATE AMINOTRANSFERASE, LOCAL LAB | 6 | 4 | 6
  ALANINE AMINOTRANSFERASE, LOCAL LAB: number analyzed (Participants) | 203 | 205 | 406
  ALANINE AMINOTRANSFERASE, LOCAL LAB | 9 | 3 | 10
  BILIRUBIN, TOTAL, LOCAL LAB: number analyzed (Participants) | 202 | 205 | 406
  BILIRUBIN, TOTAL, LOCAL LAB | 0 | 1 | 0
  CREATININE, LOCAL LAB | 4 | 0 | 3
  HYPERNATREMIA: number analyzed (Participants) | 203 | 204 | 406
  HYPERNATREMIA | 0 | 0 | 0
  HYPONATREMIA: number analyzed (Participants) | 203 | 204 | 406
  HYPONATREMIA | 12 | 1 | 13
  HYPERKALEMIA | 1 | 2 | 4
  HYPOKALEMIA | 1 | 2 | 2
  HYPERCALCEMIA: number analyzed (Participants) | 199 | 199 | 397
  HYPERCALCEMIA | 1 | 0 | 1
  HYPOCALCEMIA: number analyzed (Participants) | 199 | 199 | 397
  HYPOCALCEMIA | 0 | 1 | 1
  HYPERMAGNESEMIA: number analyzed (Participants) | 198 | 203 | 405
  HYPERMAGNESEMIA | 3 | 2 | 3
  HYPOMAGNESEMIA: number analyzed (Participants) | 198 | 203 | 405
  HYPOMAGNESEMIA | 0 | 1 | 1
  HYPERGLYCEMIA: number analyzed (Participants) | 99 | 109 | 211
  HYPERGLYCEMIA | 3 | 1 | 4
  HYPOGLYCEMIA: number analyzed (Participants) | 199 | 195 | 402
  HYPOGLYCEMIA | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from a participants first dose to their study completion (up to approximately 72 months) SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 50 weeks).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication. Prespecified to be collected with Parts A and B combined in the Nivo + Ipi and Placebo treatment strategies.
Groups:
- Treatment Part A and B: Nivo + Ipi: Nivolumab 240 mg every 2 weeks and ipilimumab 1 mg/kg every 6 weeks (or every third nivolumab dose if dosing is delayed).
- Treatment Part A and B: Placebo: Placebo infusions at the same frequency of nivolumab and ipilimumab infusions.
Arm/Group | Treatment Part A and B: Nivo + Ipi | Treatment Part A and B: Placebo | Treatment Part B: Nivo
All-Cause Mortality (participants affected / at risk) | 65/611 | 55/619 | 22/411
Serious Adverse Events (participants affected / at risk) | 196/608 | 49/614 | 56/408
Other Adverse Events (participants affected / at risk) | 544/608 | 469/614 | 325/408
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Part A and B: Nivo + Ipi (N=608) | Treatment Part A and B: Placebo (N=614) | Treatment Part B: Nivo (N=408)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Myocardial injury (Cardiac disorders) | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 3 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Paraduodenal hernia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 21 | 0 | 3
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 0
Hypophysitis (Endocrine disorders) | 12 | 0 | 0
Hypopituitarism (Endocrine disorders) | 4 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0 | 0
Lymphocytic hypophysitis (Endocrine disorders) | 1 | 0 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 2 | 0 | 0
Thyroiditis (Endocrine disorders) | 2 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1
Orbital myositis (Eye disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0
Serous retinal detachment (Eye disorders) | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0
Autoimmune colitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 12 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 16 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 6 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Mesenteric panniculitis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Disease recurrence (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 2 | 0 | 0
Malaise (General disorders) | 1 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 4 | 0 | 1
Sudden death (General disorders) | 1 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 2 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 | 0 | 1
Subacute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Sarcoidosis (Immune system disorders) | 2 | 0 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 1
COVID-19 (Infections and infestations) | 1 | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Encephalitis (Infections and infestations) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0
Gastrointestinal fungal infection (Infections and infestations) | 1 | 0 | 0
Hepatitis E (Infections and infestations) | 0 | 1 | 0
Herpes zoster meningitis (Infections and infestations) | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0
Meningitis aseptic (Infections and infestations) | 2 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 6 | 1 | 1
Postoperative wound infection (Infections and infestations) | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 2 | 1
Septic shock (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 0 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0
Open fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Splenic injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0
General physical condition abnormal (Investigations) | 1 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 | 0 | 3
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0 | 3
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 0 | 2
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 4 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 2
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Encephalitis autoimmune (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Immune-mediated encephalitis (Nervous system disorders) | 2 | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Neurological decompensation (Nervous system disorders) | 0 | 1 | 0
Osmotic demyelination syndrome (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Tension headache (Nervous system disorders) | 1 | 0 | 0
Device breakage (Product Issues) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 13 | 1 | 2
Bladder hypertrophy (Renal and urinary disorders) | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1
Immune-mediated nephritis (Renal and urinary disorders) | 1 | 0 | 0
Nephritis (Renal and urinary disorders) | 1 | 0 | 1
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Assisted suicide (Surgical and medical procedures) | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Part A and B: Nivo + Ipi (N=608) | Treatment Part A and B: Placebo (N=614) | Treatment Part B: Nivo (N=408)
Anaemia (Blood and lymphatic system disorders) | 42 | 24 | 21
Adrenal insufficiency (Endocrine disorders) | 52 | 4 | 13
Hyperthyroidism (Endocrine disorders) | 98 | 8 | 47
Hypothyroidism (Endocrine disorders) | 131 | 28 | 54
Abdominal pain (Gastrointestinal disorders) | 40 | 44 | 21
Constipation (Gastrointestinal disorders) | 57 | 49 | 29
Diarrhoea (Gastrointestinal disorders) | 180 | 120 | 77
Dry mouth (Gastrointestinal disorders) | 49 | 15 | 20
Nausea (Gastrointestinal disorders) | 102 | 73 | 53
Vomiting (Gastrointestinal disorders) | 52 | 30 | 27
Asthenia (General disorders) | 72 | 55 | 46
Fatigue (General disorders) | 189 | 158 | 99
Pyrexia (General disorders) | 61 | 25 | 13
COVID-19 (Infections and infestations) | 15 | 19 | 29
Alanine aminotransferase increased (Investigations) | 74 | 24 | 34
Aspartate aminotransferase increased (Investigations) | 60 | 15 | 22
Blood creatinine increased (Investigations) | 82 | 59 | 40
Decreased appetite (Metabolism and nutrition disorders) | 71 | 19 | 15
Hyperglycaemia (Metabolism and nutrition disorders) | 35 | 25 | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 111 | 97 | 58
Back pain (Musculoskeletal and connective tissue disorders) | 45 | 66 | 48
Myalgia (Musculoskeletal and connective tissue disorders) | 57 | 47 | 39
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 29 | 22
Dizziness (Nervous system disorders) | 37 | 38 | 17
Headache (Nervous system disorders) | 102 | 89 | 53
Insomnia (Psychiatric disorders) | 51 | 37 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 66 | 67 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 36 | 38 | 21
Dry skin (Skin and subcutaneous tissue disorders) | 47 | 30 | 19
Pruritus (Skin and subcutaneous tissue disorders) | 213 | 103 | 103
Rash (Skin and subcutaneous tissue disorders) | 131 | 57 | 50
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 51 | 6 | 23
Hypertension (Vascular disorders) | 31 | 45 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT03138512/Prot_SAP_000.pdf